CLINICAL TRIAL: NCT07101549
Title: A Single-center, Single-arm, Dose-escalation Exploratory Clinical Trial on the Safety, Efficacy, and Pharmacokinetics of R-Star001 Cell Injection in Patients With Nectin-4-positive Advanced Solid Tumors
Brief Title: Treating Nectin-4-positive Advanced Solid Tumors With R-Star001 (Nectin-4-CART-IL18)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: changjianhua (Other)
Responsible Party: Sponsor-Investigator, changjianhua, Professor, Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center
Organization: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YW2024-42-3
Record Dates: First submitted 2025-07-17; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
Keywords: Nectin-4-positive advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nectin-4-targeted CAR T-cell injection with inducing IL-18 secretion (Experimental): Experimental: Phase 1, open-label, single-arm trial. Drug: Nectin-4-targeted CAR T-cell injection with inducing IL-18 secretion.
  Interventions: Drug: R-Star001

INTERVENTIONS:
Drug: R-Star001 — Drug: Nectin-4-targeted CAR T-cell injection with inducing IL-18 secretion (R-Star001).
  The trial consists of a traditional '3 + 3' pattern dose-escalation phase and a dose-expansion phase.

SUMMARY:
A single-center, single-arm, dose-escalation exploratory clinical trial on the safety, efficacy, and pharmacokinetics of R-Star001 cell injection in patients with Nectin-4-positive advanced solid tumors.

DETAILED DESCRIPTION:
This study is a prospective, single-center, single-arm, open-label, single-dose administration dose-finding study, which aims to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor efficacy characteristics of the R-Star001 cell injection in subjects with Nectin-4 positive advanced solid tumors.

The study will enroll subjects with pathologically confirmed advanced solid tumors (including, but not limited to breast cancer, urothelial carcinoma, colorectal cancer, head and neck squamous cell carcinoma, ovarian cancer, esophageal cancer, lung cancer) who have failed standard therapy; AND immunohistochemical analysis of histological or cytological tumor specimens demonstrates moderate to high Nectin-4 expression.

This prospective, single-center, single-arm, open-label study employs a single-dose administration design across two sequential stages. Stage 1 (Dose Escalation) utilizes an accelerated titration approach with standard '3+3' dose escalation to evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of R-Star001 Cell Injection in subjects with Nectin-4 positive advanced solid tumors, thereby determining expansion dose levels based on integrated cohort data. Stage 2 (Dose Expansion) will enroll up to 9 subjects per cohort (including escalation-phase subjects) at 1-2 selected dose levels to further characterize safety and efficacy. The Recommended Phase II Dose (RP2D) will be determined post-infusion through comprehensive analysis of Stage 1 safety/efficacy outcomes, pharmacokinetic profiles, and prior preclinical/clinical evidence.

Main purpose:

the safety and tolerability of R-Star001 cell injection in patients with Nectin-4 positive advanced solid tumors, and determine the Recommended Phase II Dose (RP2D).

Secondary Purpose:

The pharmacokinetic and pharmacodynamic characteristics of R-Star001 cell injection in patients with Nectin-4 positive advanced solid tumors; To preliminarily evaluate the efficacy of R-Star001 cell injection in patients with Nectin-4 positive advanced solid tumors.

Evaluate the immunogenicity of R-Star001 cell injection.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical trial; fully understand and be informed about this study and sign the informed consent form; be willing to follow and be able to complete all trial procedures;
2. At the time of screening, the age should be between 18 and 70 years old (inclusive), regardless of gender;
3. Patients with pathologically diagnosed advanced solid tumors (including but not limited to breast cancer, urothelial cancer, colorectal cancer, head and neck squamous cell carcinoma, ovarian cancer, esophageal cancer, pancreatic cancer, non-small cell lung cancer (NSCLC)) who have failed standard treatment;
4. The histological or cytological tumor specimens have been confirmed by immunohistochemistry to have high or moderate expression of Nectin-4;
5. The patient has at least one measurable lesion (according to the requirements of RECIST version 1.1, the long diameter of the measurable lesion on spiral CT scan is ≥ 10mm or the short diameter of the enlarged lymph node is ≥ 15mm. See Annex 1 for RECIST version 1.1);
6. At the time of enrollment, the expected survival time is more than 12 weeks;
7. At the time of screening, the laboratory tests should meet the following requirements:

   * White blood cell count ≥ 3.0×10⁹/L;
   * Neutrophil count ≥ 1.5×10⁹/L;
   * Lymphocyte count ≥ 0.5×10⁹/L;
   * Hemoglobin ≥ 90 g/L;
   * Platelets ≥ 75×10⁹/L;
   * Serum total bilirubin ≤ 2.0× the upper limit of normal value (ULN);
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN; For patients with liver metastases or those with primary liver tumor lesions, the aspartate transaminase and alanine transaminase should be ≤ 5×ULN. For patients with a history of Gilbert's syndrome/suspected of having the disease, the total bilirubin (TBIL) should be ≤ 3×ULN;
   * Creatinine < 1.5×ULN and endogenous creatinine clearance rate ≥ 50 mL/minute (Cockcroft-Gault method for calculating creatinine clearance rate: For men, creatinine clearance rate = [(140 - age) × body weight (kg)] / [0.818 × creatinine (μmol/L)]; For women, creatinine clearance rate = [(140 - age) × body weight (kg) × 0.85] / [0.818 × creatinine (μmol/L)]).
8. Good lung function, with a baseline fingertip pulse oximetry saturation ≥ 95% in an indoor air environment;
9. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0 or 1;
10. Female subjects with reproductive potential must undergo a serum pregnancy test at the time of screening and before receiving pre-treatment, and the result must be negative. They should be willing to use a highly effective and reliable contraceptive method within 1 year after the last use of the test drug. Available methods include: bilateral tubal ligation/bilateral salpingectomy or bilateral fallopian tube occlusion; or approved oral, injectable or implanted hormonal contraceptive methods; or barrier contraceptive methods: condoms or occlusive caps (diaphragm or cervical/vaginal vault caps) containing spermicidal foam/gel/membrane/cream/suppository;
11. For men who have an active sexual life with women of reproductive potential and have not had a vasectomy, they must agree to use a barrier method of contraception, such as a condom containing spermicidal foam/gel/membrane/cream/suppository, or their spouses should use a contraceptive method (see Inclusion Criteria item 10). Moreover, all men are absolutely prohibited from donating sperm within 1 year after receiving the last infusion of the test drug;
12. A venous access can be established, and the collection of peripheral blood mononuclear cells can be carried out as judged by the investigator.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Those with a history of allergy to immunotherapy, allergy to related drugs, a history of severe allergies in the past, and allergy to the components of R-Star001;
3. Patients with other malignant tumors, except for the following situations: cured non-melanoma skin cancer, in-situ cervical cancer, localized prostate cancer, superficial bladder cancer, and other malignant tumors with a disease-free survival period of more than 3 years;
4. Symptomatic intracranial or spinal cord metastasis of the tumor;
5. Positive for hepatitis B surface antigen (HBsAg) positive, hepatitis B e-antigen (HBeAg) positive, hepatitis B e-antibody (HBeAb) positive, hepatitis B core antibody (HBcAb) positive, hepatitis C virus antibody (HCV-Ab) positive, anti-Treponema pallidum antibody (TP-Ab) ; subjects meeting any one of the above items;
6. Any uncontrolled active infection, including but not limited to active tuberculosis and other bacterial, viral or fungal infections requiring drug treatment. Subjects who are using drugs to prevent infection can continue the trial as judged by the investigator;
7. Those who have received live vaccines or live attenuated vaccines within 4 weeks before apheresis;Have received the last dose of antitumor therapy (chemotherapy, endocrine therapy, immunotherapy, targeted therapy, tumor embolization, or Chinese herbal medicine with antitumor indications, etc.) within 3 weeks before leukocyte apheresis;
8. The toxic and side effects caused by previous treatment have not recovered to CTCAE ≤ Grade 1;
9. Those who have received any genetically engineered modified cell therapy in the past;
10. Subjects at high risk of causing bleeding or perforation;
11. Subjects who require anticoagulant therapy;
12. Subjects who require long-term antiplatelet therapy;
13. Subjects with a history of organ transplantation or those waiting for organ transplantation;
14. Subjects who have undergone major surgery or suffered significant trauma within 4 weeks, or those who are expected to undergo major surgery during the study period;
15. Those with other serious diseases that may limit the subject's participation in this trial;
16. Subjects with signs of central nervous system diseases or clinically significant abnormal results of neurological examinations;
17. Those with a history of abuse of psychotropic drugs who are unable to quit or those with a history of mental disorders;
18. Subjects who, as evaluated by the investigator, are unable or unwilling to comply with the requirements of the study protocol;
19. Situations in which the subject, as judged by the investigator, is not suitable for the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days of single infusion
  Dose limiting toxicity (DLT) in the dose escalation phase
Adverse events (AEs) | 1 year
  The incidence rate of treatment-emergent adverse events (TEAEs), the incidence rate of treatment-related adverse events, and the incidence rate of adverse events of special interest (AESIs)
Maximum tolerated dose (MTD) | 28 days of single infusion
  Maximum tolerated dose (MTD) in the dose escalation phase

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year
  After treatment with R-Star001 cell infusion, the proportion of subjects whose tumors achieved complete response (CR) or partial response (PR). The objective response rate of tumors is only calculated for patients with measurable diseases according to the RECIST 1.1 criteria.
Disease Control Rate (DCR) | 1 year
  After treatment with R-Star001 cell infusion, the proportion of subjects who achieved complete response, partial response, and stable disease.
Progression - free survival (PFS) | 1 year
  The time from the date of starting the treatment with R-Star001 cell infusion to the date of the first radiological confirmation of disease progression (PD) or the date of death (due to any cause), whichever occurs first.
Overall survival (OS) | 1 year
  The time from the date of starting the treatment with R-Star001 cell infusion to the date of death (caused by any reason).
Immunogenicity | 1 year
  The incidence of antibodies against the R-Star001 cell injection and the titer of positive samples.
Cellular pharmacokinetics (Cmax) | 1 year
  The peak concentration (Cmax)of CAR copy number in peripheral blood for R-Star001 cell injection.
Cellular pharmacokinetics (Tmax) | 1 year
  Time to peak concentration (Tmax) of CAR copy number in peripheral blood for R-Star001 cell injection.
Cellular pharmacokinetics (AUC) | 1 year
  Area under the plasma concentration-time curve (AUC) of R-Star001 cell injection in peripheral blood over 28/90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Chang, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center
Locations (1):
- Cancer Hospital Chinese Academy Of Medical Sciences,Shenzhen Center, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No